CLINICAL TRIAL: NCT06995768
Title: Normative Data for Sweating Rate, Sweat Sodium Concentration and Sweat Sodium Loss in Female Athlete
Status: Recruiting | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2506
Record Dates: First submitted 2025-04-30; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sweat Rate
Keywords: sweat; sodium loss; sweat patch; athlete; healthy volunteer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female team sports athletes aged 13 and over: Multiple athletic teams at locations in USA and UK
  Interventions: Other: Sweat patch

INTERVENTIONS:
Other: Sweat patch — Wear sweat patch during regular team sports practice session

SUMMARY:
The main objectives are to determine sweat sodium concentration [Na+], whole body sweat rate (WBSR) and rate of sweat sodium loss (RSSL) in female athletes aged 13 and above during their normal planned training session across various sports (basketball, soccer, volleyball, cheer, flag football and softball).

DETAILED DESCRIPTION:
The testing procedures will follow the standardized Gatorade Sports Sciences GSSI sweat testing protocol using the absorbent sweat patch technique, to measure local sweat [Na+], which will be normalized to whole-body sweat [Na+]. Whole-body sweat rate (WBSR) will be calculated based on changes in exercise body mass, pre to post training, and adjusted for food and fluid intake, as well as urine and stool loss. The rate of sweat sodium loss (RSSL) will be determined as the product of sweat [Na+] and WBSR.

Secondary outcomes are pre-exercise hydration status measured by urine specific gravity (USG) and estimation of menstrual cycle phase collected by self-report date of last menstrual cycle.

Athletes will complete a single day of testing, unless a repeat test is requested by the team's performance staff. In this case, athletes will undergo the exact same protocol as described above.

ELIGIBILITY:
Inclusion Criteria:

Subject is female

* Subject is 13yrs+
* Subject has been cleared for sport participation by their personal or team physician and/or coach-led practice/training.
* Subject is participating in sport on the youth/ amateur/ collegiate/professional/elite level
* If under 18, a parental/guardian consent form will be completed.

Exclusion Criteria:

* As this study is undertaken at the athletes training facility, the medical staff at the team/club will advise on who should/ should not take part.
* Subject has an allergy to adhesives (e.g., experiences rash reactions to typical adhesive bandages

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Reason female only is lack of sports science sweat research data specific to female athletes
Study Population: Healthy female athletes in coach-led team sports
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Regional sweat [Na+] | One day from start through end of a single coach-led normal training practice session. Practice duration will be dictated by coaching staff.
  Absorbent patch technique (3M TegadermTM + Pad; 3M, St. Paul, MN; pad size 10 cm2 with an absorbent capacity of ~1.3 g) to left and right dorsal arm. An additional patch on the right scapula may be added depending on the accessibility to the sites on the body and the nature of the sport. Analyzed using a HORIBA (LAQUAtwin Na-11)
Whole body sweat rate (WBSR) WBSR | One day from start through end of a single coach-led training normal training practice session. Practice duration will be dictated by coaching staff.A
  Pre- versus post body mass on scale, taking into account food and fluid intake, urine and stool output
Rate of sweat sodium loss (RSSL) | One day from start through end of a single coach-led normal training practice session. Duration will be dictated by coaching staff.
  The rate of sodium sweat loss (RSSL) will be determined as the product of sweat [Na+] and whole-body sweat rate (WBSR)

SECONDARY OUTCOMES:
Urine specific gravity (USG) | Pre-exercise at one coach-led normal training practice session.
  Unit not applicable
Fluid intake | One day from start through end of a single coach-led normal training practice session. Duration will be dictated by coaching staff.
  Weighing pre-filled bottles before and after exercise, beverage choice of water, and Gatorade, or G2
Carbohydrate intake | One day from start through end of a single coach-led normal training practice session. Duration will be dictated by coaching staff.
  Grams of carbohydrate consumed through food and beverages

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Randell, PhD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- Gatorade Sports Science Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No